CLINICAL TRIAL: NCT05839938
Title: The Role of Vitamin D in Corneal Epithelial Barrier Function, Ocular Microbiome, Ocular Inflammation, and Visual Acuity of Children With Allergic Conjunctivitis
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CMUH111-REC1-044
Record Dates: First submitted 2023-04-21; First posted 2023-05-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Allergic Conjunctivitis
Keywords: allergic conjunctivitis, immune privilege; corneal epithelial barrier; microbiota; vitamin D; ocular microenvironment; visual acuity; vitamin D receptor gene polymorphism; ocular surface and intraocular inflammation
MeSH Terms: conditions — Conjunctivitis, Allergic; Uveitis | interventions — Vitamin D

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): Vitamin D (2000IU/day) for 6 months
  Interventions: Other: Vitamin D
- Control group (Placebo Comparator): placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Vitamin D — Vitamin D (2000IU/day) for 6 months
  Arms: Treatment group
Other: Placebo — Placebo
  Arms: Control group

SUMMARY:
A double-blind study to evaluate the role of vitamin D in corneal epithelial barrier function, ocular microbiome, ocular inflammation, and visual acuity of children with allergic conjunctivitis.

DETAILED DESCRIPTION:
The prevalence of allergic conjunctivitis (AC) has rapidly increased in recent decades, resulting in a significant global public health concern. The ocular surface is a unique mucosal immune compartment in which immunological features act in concert to foster a tolerant microenvironment (immune privilege). The corneal epithelial barrier is the first line of defense that forms a protective barrier against pathogens, pollutants, and allergens. The ocular microbiota has a role in maintaining the homeostasis of the ocular surface and preservation of barrier function. Vitamin D functions as enforcing intercellular junctions and maintaining intestinal epithelial barrier integrity; metabolites from the gut microbiota may also regulate expression of vitamin D receptor (VDR). Low serum vitamin D levels have been shown to predispose to a variety of allergic disorders. A recent study shows that corneas contain vitamin D and VDR; vitamin D enhances corneal epithelial barrier function. However, research data of the role of vitamin D in ocular microenvironment of AC are insufficient and controversial. In recent research, the investigators found allergic inflammation of ocular surface weakened corneal epithelial barrier, modulated the signal pathway of retinal pigment epithelial cells, and enhanced scleral tissue remodeling, resulting in myopia in progression. However, there are few studies available to investigate the role of vitamin D in ocular surface microenvironment, ocular inflammation, and visual acuity in AC. Moreover, understanding the interaction of vitamin D, ocular microbiota, and ocular inflammation may provide a new target for the development of therapeutic interventions of ocular allergy and restore visual function.

ELIGIBILITY:
Inclusion Criteria:

1. Children aged 6-18 years with allergic conjunctivitis (AC) diagnosed by ophthalmologists or allergists

Exclusion Criteria:

1. Previous eye surgery
2. Active eye infection
3. Any active inflammatory eye disease except AC
4. Systemic steroid use within 28 days of study

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-08-08 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Levels of vitamin D | Month 0
  Vitamin D will be measured in a blood sample by ELISA to determine baseline status.
Levels of vitamin D | Month 6
  Vitamin D will be measured in a blood sample to follow the change from baseline in vitamin D level at month 6.
Single nucleotide polymorphism of vitamin D receptor and vitamin D binding protein | Month 0
  Single nucleotide polymorphism (SNP) genotyping will be performed in a blood sample by using TaqMan SNP genotyping assays.
Microbiome | Month 0
  Nasal, subconjunctival and anal swabs will be used to detect ocular surface, nasal and intestinal microbiome by using 16S rRNA sequencing to determine baseline status.
Microbiome | Month 6
  Nasal, subconjunctival and anal swabs will be used to detect ocular surface, nasal and intestinal microbiome by using 16S rRNA sequencing, and to follow the change from baseline in microbiome at month 6.
Total IgE | Month 0
  Plasma total IgE concentration will be measured by microparticle immunoassay (IMx analyzer, Abbott Laboratories, Abbott Park, IL) and ELISA to determine baseline status.
Total IgE | Month 6
  Plasma total IgE concentration will be measured by microparticle immunoassay (IMx analyzer, Abbott Laboratories, Abbott Park, IL) and ELISA to follow the change from baseline in total IgE at month 6.
Allergen-specific IgE | Month 0
  Plasma allergen-specific IgE will be measured by BioIC ®.

SECONDARY OUTCOMES:
mini-Rhinoconjunctivitis Quality of Life Questionnaire (mini-RQLQ) | Month 0 to Month 6
  mini-RQLQ is to measure a the level of severity of a set of symptoms of functional impairments due to rhinoconjunctivitis. 14 questions each range 0-6 (6 is most severe). Total range 0-84 (higher scores reflect lower quality of life.)

CONTACTS AND LOCATIONS:
Locations (1):
- China Medical University Hospital, Taichung, Taiwan